CLINICAL TRIAL: NCT03840109
Title: Emotional Support Messages Following a Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: San Diego State University (Other); University of Arizona (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-19957
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Psychological Stress; Anxiety
Keywords: emotional support; cancer
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All participants will take an online questionnaire which includes their evaluation of one of 18 different emotional support messages randomly assigned through the Qualtrics survey system. The participants answer a series of closed ended scales regarding quality of the support message, supporter's competence, amount of emotional improvement they experienced after reading the message, and likelihood to seek support from the person writing the message.
  Interventions: Behavioral: Questionnaire 1a; Behavioral: Questionnaire 1b; Behavioral: Questionnaire 2a; Behavioral: Questionnaire 2b; Behavioral: Questionnaire 3a; Behavioral: Questionnaire 3b; Behavioral: Questionnaire 4a; Behavioral: Questionnaire 4b

INTERVENTIONS:
Behavioral: Questionnaire 1a — Participants will be randomly shown two versions of messages in which the last 20% of the message consists of negative statements of criticism and rate of the effectiveness of the message.
Behavioral: Questionnaire 1b — Participants will be randomly shown two versions of messages in which the first 20% of the message consists of negative statements of criticism and rate of the effectiveness of the message.
Behavioral: Questionnaire 2a — Participants will be randomly shown two versions of messages in which the last 40% of the message consists of negative statements of criticism and rate of the effectiveness of the message.
Behavioral: Questionnaire 2b — Participants will be randomly shown two versions of messages in which the first 40% of the message consists of negative statements of criticism and rate of the effectiveness of the message.
Behavioral: Questionnaire 3a — Participants will be randomly shown two versions of messages in which the last 60% of the message consists of negative statements of criticism and rate of the effectiveness of the message.
Behavioral: Questionnaire 3b — Participants will be randomly shown two versions of messages in which the first 60% of the message consists of negative statements of criticism and rate of the effectiveness of the message.
Behavioral: Questionnaire 4a — Participants will be randomly shown two versions of messages in which the last 80% of the message consists of negative statements of criticism and rate of the effectiveness of the message.
Behavioral: Questionnaire 4b — Participants will be randomly shown two versions of messages in which the first 80% of the message consists of negative statements of criticism and rate of the effectiveness of the message.

SUMMARY:
Cancer patients will be randomly shown one of 18 emotional support messages created by the research team that differ based on how much of the message consists of positive statements and how much consists of negative statements. The messages with negative statements also differ based on whether the negative statements occur at the start or end of the message. After viewing the message, participants have the opportunity to rate the effectiveness of the message, to what extent the message made them feel better, and to what extent the message affects how they view the message provider as a useful source of emotional support.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants with a diagnosis of breast, prostate, thoracic or digestive cancer in the past 3 years
* Participants consented to Moffitt's Total Cancer Care (TCC) protocol and indicating a willingness to be contacted for future research by including an email contact.
* Ability to read and write fluently in English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients
Sampling Method: Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Message Effectiveness Scale | Through study completion, up to 1 year
  Perceptions of message effectiveness will be tested through 4 ANOVA models that will test for differences between participants who received different messages in terms of perceived message effectiveness.
Affective Improvement Scale | Through study completion, up to 1 year
  Perceptions of message effectiveness will be tested through 4 ANOVA models that will test for differences between participants who received different messages in terms of self-reports of emotional improvement.

SECONDARY OUTCOMES:
Supporter Competence Scale | Through study completion, up to 1 year
  Perceptions of message effectiveness will be tested through 4 ANOVA models that will test for differences between participants who received different messages in terms of perceptions of supporter competence.
Likelihood of Seeking Support Scale | Through study completion, up to 1 year
  Perceptions of message effectiveness will be tested through 4 ANOVA models that will test for differences between participants who received different messages in terms of their likelihood to seek support from the supporter in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Maija Reblin, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03840109/Prot_SAP_000.pdf